CLINICAL TRIAL: NCT00336934
Title: A Randomized, Double-Blind, Placebo-Controlled Study of The Effects of Pomegranate Extract On Rising Prostate-Specific Antigen Levels In Men Following Primary Therapy
Brief Title: Pomegranate Extract in Treating Patients With Rising Prostate-Specific Antigen Levels After Surgery or Radiation Therapy for Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roll International Corporation (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: MaryBethAudickas, Radiant Research - Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000480402; P30CA016042 (NIH); ROLL-GUP-0205-1; UCLA-0507059-01; NCT00413530 (obsolete NCT alias)
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral pomegranate extract daily.
  Interventions: Dietary Supplement: pomegranate juice
- Arm II (Placebo Comparator): Patients receive oral placebo daily.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: pomegranate juice — Given orally daily.
  Arms: Arm I
Other: placebo — Given orally daily.
  Arms: Arm II

SUMMARY:
RATIONALE: Pomegranate extract may keep prostate cancer from growing in patients with rising prostate-specific antigen (PSA) levels after surgery or radiation therapy for localized prostate cancer.

PURPOSE: This randomized trial is studying how well pomegranate extract works in treating patients with rising PSA levels after surgery or radiation therapy for localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effects of pomegranate extract in patients with and rising prostate-specific antigen (PSA) levels after surgery or radiotherapy for localized prostate cancer.
* Determine the effect of a daily oral dose of pomegranate extract on the absolute value of PSA and on the change in PSA doubling time in these patients.

Secondary

* Assess toxicities associated with daily oral dosing of pomegranate extract in these patients.
* Determine the effect of pomegranate extract on positive PSA doubling-time outcome, defined as greater than 150% baseline or a negative post-treatment PSA doubling time (i.e., declining PSA).

OUTLINE: This is a multicenter, double-blind, placebo-controlled, randomized study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral pomegranate extract daily.
* Arm II: Patients receive oral placebo daily. Treatment in both arms continues for up to 1 year in the absence of disease progression.

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Must have completed prior surgery, cryotherapy, or radiotherapy for the primary tumor
* Documented rising prostate-specific antigen (PSA)

  * Absolute level of PSA > 0.2 ng/mL after surgery
  * Absolute level of PSA > 1.0 ng/mL after radiation or cryotherapy
  * Absolute level of PSA ≥ 0.4 ng/mL after multiple treatment modalities (e.g., surgery with radiotherapy or radiotherapy with cryotherapy)
  * PSA must be ≥ 100% above best nadir achieved
  * PSA doubling time > 3 months or ≤ 24 months

    * Patients must have ≥ 3 rising PSA time points above the minimum nadir achieved over ≥ 6 months

      * The interval between PSA time points must be > 2 weeks
* PSA ≤ 7.0 ng/mL
* Patients who underwent radical prostatectomy and never achieved undetectable serum PSA after surgery are not eligible
* Gleason score ≤ 7
* No histologically positive lymph nodes
* No evidence of metastatic disease by physical examination, CT scan, or bone scan

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* ECOG performance status 0 or 1
* No significant concomitant medical or psychiatric conditions that would limit study compliance
* No known allergies to pomegranate extract
* No known diabetes with hemoglobin A_1c level > 7.0% in the past 3 months

  * Diabetic patients entering study who have not had hemoglobin A_1c level measured in the past 3 months must have levels measured at study initiation
* No clinically abnormal laboratory values > 2 times the upper limit of normal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior and no concurrent experimental drugs, high-dose steroids, or other cancer treatment
* No hormonal therapy, with the exception of neoadjuvant androgen-deprivation therapy (ADT), prior to or concurrent with primary therapy

  * Patients who received prior neoadjuvant ADT must have serum testosterone ≥ 150 ng/dL
* No prior or concurrent hormonal therapy for rising PSA after primary therapy for prostate cancer
* No finasteride or dutasteride at any time point after primary therapy and during study therapy
* No other concurrent commercial pomegranate products
* No other concurrent systemic or local therapy for prostate cancer
* Concurrent dietary/herbal supplements (e.g., saw palmetto or selenium) allowed provided dose has been stable for ≥ 2 months prior to study entry and there are no plans to change or stop the supplements during study therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-11; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Objective response | 12 months

SECONDARY OUTCOMES:
Response duration | 12 months
Effects of pomegranate extract on prostate-specific antigen (PSA) doubling and velocity times | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Pantuck, MD, Principal Investigator — Jonsson Comprehensive Cancer Center; Arie Belldegrun, MD, FACS, Principal Investigator — Jonsson Comprehensive Cancer Center